CLINICAL TRIAL: NCT01905761
Title: UMP Lifestyle Medicine Program
Status: Withdrawn | Type: Observational
Why Stopped: Project abandoned
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: UMP Lifestyle Medicine Program
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Obesity
Keywords: obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To systematically follow patients seen at the University of Minnesota's Lifestyle Medicine Program for Weight Management.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen who sign medical release form

Exclusion Criteria:

None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are adults with obesity (BMI > 30) seen at our Lifestyle Medicine program in weight management at the University of Minnesota
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Body weight change | 3 - 60 months
  Body weight change from clinical program entry until discharge

SECONDARY OUTCOMES:
Body fat percentage | 3-60 months
  Assess body fat percentage change from clinical program entry until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Steven Stovitz, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota's Smiley's clinic, Minneapolis, Minnesota, United States